CLINICAL TRIAL: NCT06873854
Title: Evaluation of a Phase II, Single-arm, Multicenter, Open-label Clinical Study on LM-108 Injection in Combination With Toripalimab for Advanced Malignant Solid Tumors in Patients With Unresectable or Metastatic Microsatellite Highly Unstable (MSI H) or Mismatch Repair Defects (dMMR) Who Have Failed Previous Treatment With Anti-PD-1/PD-L1 Drugs
Brief Title: A Study of LM-108 in Combination With Toripalimab in Subjects With Advanced Solid Tumours
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: LaNova Medicines Limited (Industry)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LM-108-II-01
Record Dates: First submitted 2025-02-13; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LM-108 in Combination with Toripalimab (Experimental)
  Interventions: Drug: LM-108; Drug: Toripalimab

INTERVENTIONS:
Drug: LM-108 — Q3W, Intravenous Drip
Drug: Toripalimab — Q3W, Intravenous Drip

SUMMARY:
Based on overall response rate (ORR) as assessed by the Independent Review Committee (IRC) against the Response Evaluation Criteria in Solid Tumors (RECIST v1.1) criteria for Solid Tumor Efficacy, To evaluate the efficacy of LM-108 in combination with Toripalimab in patients with advanced malignant solid tumours with unresectable or metastatic MSI-H/dMMR who have failed previous anti-PD-1 /PD-L1 therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with advanced solid tumors diagnosed by pathology have evidence of advanced stage or metastasis that cannot be surgically removed. And the MSI-H status will be confirmed by central laboratory designated of the sponsor.
2. Aged 18.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
4. At least one measurable lesion.
5. Subjects who have failed previous monotherapy with anti-PD-1/PD-L1 drugs or combination (synchronous or sequential) with other systemic treatments and unresectable or metastatic late stage MSI-H/dMMR solid tumors.
6. Subjects must have Archived Samples or fresh tumor tissue specimens are required for testing.
7. Any adverse event from prior anti-tumor therapy and surgery has recovered to ≤ grade 1 of CTCAE v5.0.
8. Subjects must show appropriate organ and marrow function in laboratory examinations.
9. Women of childbearing potential (WOCBP) and Male participants must agree to use one medically recognized contraceptive measures of contraception, during the study and for 6 months after the last dose of study drug.
10. Subjects who are willing to participate in the study and sign the informed consent form (ICF) prior to any procedure.

Exclusion Criteria:

1. Subjects with symptomatic/active central nervous system (CNS) metastases.
2. Subject who have uncontrollable pleural effusion, pericardial effusion, and ascites despite treatment such as puncture and drainage Within 14 days prior to enrollment; Pericardial effusion accompanied by clinical symptoms or moderate or above.
3. Subjects' weight decreased by more than 20% within the first 2 months of enrollment.
4. Poorly controlled tumor-related pain.
5. Subjects who received anti-tumour treatment, , major surgery, immunosuppressive drugs and live attenuated vaccines before enrollment.
6. Subjects have received anti-tumor immunotherapy and experienced ≥ grade 3 immune related adverse events (irAE) or ≥ grade 2 immune related myocarditis.
7. Subjects who have other cancers within 5 years prior to entering the research.
8. Previous or current known autoimmune disease.
9. Within the first 3 months of enrollment, there have been significant clinical bleeding symptoms or clear bleeding tendencies; Arterial/venous thrombotic events that occurred within the first 6 months of enrollment.
10. Present peripheral neuropathy of grade>1 .
11. Subjects who have a history of gastrointestinal perforation and/or gastrointestinal fistula within the 6 months prior to enrollment.
12. Subjects who have been clinical signs or symptoms of intestinal obstruction and/or gastrointestinal obstruction Within 6 months prior to starting the study treatment.
13. Presence of interstitial lung disease, non infectious pneumonia, or uncontrolled systemic diseases.
14. Known to be allergic to the investigational drug or any of its excipients; Or have experienced severe allergic reactions to other monoclonal antibodies.
15. HIV infection, active HBV or HCV infection.
16. Subject who have clinical symptoms or diseases of the heart that have not been well controlled.
17. Subjects who take Systemic use of antibiotics for more than 7 days within the first 4 weeks prior to enrollment, or unexplained fever>38.5 ° C during screening/before first administration .
18. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
19. Subjects who have participated in any other drug clinical studies within 4 weeks prior to enrollment, or have not exceeded 5 half lives since the last study medication.
20. Known history of abuse or drug use of psychotropic substances.
21. Subjects who have other serious physical or mental illnesses or laboratory abnormalities and judged as not eligible to participate in this study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-03-26 (Estimated); Primary Completion 2028-01-26 (Estimated); Study Completion 2030-01-26 (Estimated)

PRIMARY OUTCOMES:
ORR | 104 weeks
  Overall Response Rate assessed by Independent Review Committee against the Response Evaluation Criteria in Solid Tumors (RECIST v1.1)

SECONDARY OUTCOMES:
AEs | 104 weeks
  Incidence of adverse events
SAEs | 104 weeks
  Incidence of serious adverse events
AE/SAE | 104 weeks
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
DOR | 104 weeks
  Duration of response assessed by Independent Review Committee against the RECIST v1.1
DCR | 104 weeks
  Disease control rate (DCR = CR + PR + SD) assessed by Independent Review Committee against the RECIST v1.1
PFS | 104 weeks
  Progression-free survival assessed by Independent Review Committee against the RECIST v1.1
Progression-free survival Rates | 104 weeks
  Independent Review Committee evaluated the Progression-free survival rates at 3 and 6 months based on RECIST v1.1
ORR | 104 weeks
  Overall Response Rate assessed by investigator against the RECIST v1.1
DOR | 104 weeks
  Duration of response assessed by investigator against the RECIST v1.1
DCR | 104 weeks
  Disease control rate (DCR = CR + PR + SD) assessed by investigator against the RECIST v1.1
PFS | 104 weeks
  Progression-free survival assessed by investigator against the RECIST v1.1
Progression-free survival Rates | 104 weeks
  Investigator evaluated the Progression-free survival rates at 3 and 6 months based on RECIST v1.1
OS | 104 weeks
  Overall survival
OS rates | 104 weeks
  Overall survival rates
Temperatures | 104 weeks
  Temperatures
Pulse in BPM | 104 weeks
  Beat per Minute
Blood Pressure | 104 weeks
  Blood Pressure in mmHg，Both systolic pressure and diastolic pressure
Weight | 104 weeks
  Weight in Kg
Height | 104 weeks
  Height in centimeter
Complete Blood Count | 104 weeks
Urine Routine test | 104 weeks
  Laboratory tests-Urine Routine test
Blood biochemistry | 104 weeks
  Laboratory tests-Blood biochemistry
Coagulation function | 104 weeks
  Laboratory tests-Coagulation function
Thyroid function | 104 weeks
  Laboratory tests-Thyroid function
Stool routine examination | 104 weeks
  Laboratory tests-Stool routine examination
Virological examination | 104 weeks
  Laboratory tests-Virological examination
Pregnancy check | 104 weeks
  Laboratory tests-Pregnancy check
LVEF | 104 weeks
  Echocardiography- LVEF(Left Ventricular Ejection Fraction) in percentage
HR | 104 weeks
  Electrocardiogram (ECG) in HR
RR | 104 weeks
  Electrocardiogram (ECG) in RR
PR | 104 weeks
  Electrocardiogram (ECG) in PR
QRS | 104 weeks
  Electrocardiogram (ECG) in QRS
QT | 104 weeks
  Electrocardiogram (ECG) in QT
QTcF | 104 weeks
  Electrocardiogram (ECG) in QTcF
ECOG score | 104 weeks
  Eastern Cooperative Oncology Group score

OTHER OUTCOMES:
iORR | 104 weeks
  Immune Overall Response Rate assessed by investigator according to the Immune Response Evaluation Criteria in solid Tumors
iDOR | 104 weeks
  Immune Duration of response assessed by investigator according to the Immune Response Evaluation Criteria in solid Tumors
iDCR | 104 weeks
  Immune Disease control rate assessed by investigator according to the Immune Response Evaluation Criteria in solid Tumors
iPFS | 104 weeks
  Immune Progression-free survival assessed by investigator according to the Immune Response Evaluation Criteria in solid Tumors
PK Parameter:Ctrough | 104 weeks
  PK Parameter:steady state at the end of the dosing interval Concentration
Immunogenicity testing | 104 weeks
  Anti-Drug antibody and Nab (if necessary) will be tested.
Biomarker correlation | 104 weeks
  For the detection of MSI or MMR, and CCR8 and PD-L1

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No